CLINICAL TRIAL: NCT01625325
Title: Medical and Psychosocial Implications of Adolescent Extreme Obesity - Acceptance and Effects of Structured Care Study, Subproject 1
Brief Title: Identification and Characterization of Youth With Extreme Obesity
Acronym: YES
Status: Completed | Type: Observational
Sponsor: Prof. Dr. Martin Wabitsch (Other)
Collaborators: University of Witten/Herdecke (Other); Charite University, Berlin, Germany (Other); University of Leipzig (Other); Universität Duisburg-Essen (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Martin Wabitsch, Division Chief Pediatric Endocrinology and Diabetology, University of Ulm
Organization: University of Ulm (Other)
Other Study IDs: U1111-1131-4384a; DRKS00004172 (Registry Identifier: Deutsches Register Klinischer Studien); 01GI1120A (Other Grant/Funding Number: Bundesministerium für Bildung und Forschung)
Record Dates: First submitted 2012-06-19; First posted 2012-06-21 (Estimated); Last update posted 2018-06-13 (Actual); Status verified 2018-06

CONDITIONS: Obesity; Extreme Obesity
Keywords: obesity, adiposity, psychosocial, healthcare, co-morbidities, low key intervention, quality of life
MeSH Terms: conditions — Obesity; Obesity, Morbid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples of fasting plasma, serum, DNA, and urine will be retained.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- extremely obese: BMI ≥35kg/m2
- obese: BMI 30-34.9kg/m2

SUMMARY:
While obese and extremely obese youth are at increased risk of health complications, especially the extremely obese group rarely seek medical care. One of the underlying reasons might be the lack of adequate treatment options. This study is a subproject of the "Medical and psychosocial implications of adolescent extreme obesity - acceptance and effects of structured care study", short: "Youth with Extreme obesity Study (YES)", which aims at improving the medical care and social support structures for youth with obesity and extreme obesity in Germany. In this subproject, information on the causes and consequences of extreme obesity will be gathered via questionnaires and medical examinations.

Obese youth and young adults (BMI ≥ 30kg/m2) between the ages of 14 and 24.9 years (initially up to 21 years) are eligible to participate. Participants will be asked to complete a series of questionnaires on their general health, psychosocial situation and wellbeing in 2-3 sessions. They will be offered a thorough medical examination comprising a general check-up, a fasting blood draw and oral glucose tolerance test, a focused orthopaedic examination, a sleep apnea screening, and an ultrasound of the liver. The aim of the study is to elicit the acceptance of diagnostic and therapeutic procedures, and to assess the frequency of co-morbidities in obese and extremely obese youth. This knowledge will optimize medical treatment and support options. Interested participants will be invited to participate in further steps of YES, which entail medical care and psycho-social support.

DETAILED DESCRIPTION:
In this multicenter study, we aim to recruit adolescents from various medical and non-medical settings and examine their acceptance of diagnostic and subsequent treatment procedures. We will compare the prevalence rates and severity of co-morbidities between adolescents with extreme obesity (BMI ≥35kg/m2)and those with less severe obesity (BMI 30-34.9kg/m2). This project is part of the "Medical and psychosocial implications of adolescent extreme obesity - acceptance and effects of structured care study", short: "Youth with extreme obesity Study (YES)", which also comprises a randomized controlled trial to investigate a novel intervention targeted at improving quality of life and social functioning of extremely obese adolescents, a structured prospective evaluation of adolescent bariatric surgery, and economic assessments of the financial burden of extreme adolescent obesity on the healthcare system.

Based on the current state of knowledge, we have formulated the following hypotheses in regards to baseline characteristics:

1. The prevalence of somatic, psychiatric and psycho-social co-morbidities is higher, and health related quality of life is lower in extremely obese youth compared to the control group.
2. The prevalence of somatic co-morbidities is equal in treatment-seeking and non treatment-seeking youth.
3. The prevalence of psychiatric co-morbidities is higher and health related quality of life is lower in treatment-seeking compared to non treatment-seeking youth.
4. The acceptance of diagnostic and therapeutic procedures is lower in extremely obese youth compared to the control group.
5. The acceptance of diagnostic and therapeutic procedures is lower in non treatment-seeking- compared to treatment-seeking youth.
6. Socio-economic status, intelligence and educational status are predictors of treatment seeking behaviour and of the acceptance of diagnostic and therapeutic procedures.

The five participating university centers are distributed across 4 geographic regions in the North (Berlin), in the West (Essen/Datteln), in the East (Leipzig) and in the South (Ulm) of Germany, and will therefore render data that are representative of Germany as a whole. We will recruit a total of 600 adolescents age 14 to 24.9 years (initial age 21 years, changed in an amendment in February 2013) with extreme obesity (BMI ≥ 35 kg/m2) and 600 adolescents with obesity (BMI 30-34.9 kg/m2) over a 24 months period. Baseline assessments include an array of standardized questionnaires and validated instruments to assess health, psycho-social situation, psychiatric co-morbidities and health related quality of life (in the amendment in February 2013, the scope of psychosocial questions was reduced), as well as a physical examination, laboratory tests, liver ultrasound, and screenings for orthopedic co-morbidities and sleep apnea. Subjects who participate in the baseline examination will be invited to participate in the subsequent components of YES.

The project will reveal comorbidity rates and psycho-social situation, and demonstrate the acceptance and outcomes of a structured healthcare program for adolescents with extreme obesity. The planned subsequent longitudinal study will provide unique information on the medical and psychosocial development of adolescents with extreme obesity in Germany.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥30kg/m2
* sufficient German language skills

Exclusion Criteria:

* none

Ages: 14 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Subjects will be recruited from the general population through different healthcare- and non healthcare settings to ascertain the inclusion of treatment-seeking and non treatment-seeking individuals. Healthcare settings include university based obesity clinics, physician offices and health insurance agencies. Non-healthcare settings include schools, job centers, and employment agencies.
Sampling Method: Non-Probability Sample
Enrollment: 429 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects that participate in the fasting blood draw | baseline
  Subjects will be offered a diagnostic blood draw. The percentage of subjects that undergo this blood draw will be calculated.

SECONDARY OUTCOMES:
Predictors of the acceptance of the diagnostic procedures | baseline
Prevalence of obesity associated psychiatric co-morbidities | baseline
  Co-morbidities will be assessed via validated patient questionnaires.
Percentage of patients that accept treatment of somatic co-morbidities | baselin
  Appropriate medical treatment of the diagnosed somatic co-morbidities will be offered to all subjects. The percentage of subjects who initiate such therapy will be calculated.
Predictors of acceptance of treatment of co-morbidities | baseline
Health related quality of life | baseline
  assessed by validated questionnaire EQ5D
Socio-economic status | baseline
  Assessed by standardized questionnaire.
Prevalence of obesity associated somatic co-morbidities | baseline
  Co-morbidities will be assessed via standardized physical examination, laboratory and apparative tests, and standardized patient questionnaires.
Percentage of patients that accept treatment of psychiatric co-morbidities | baseline
  Appropriate medical treatment of the diagnosed psychiatric co-morbidities will be offered to all subjects. The percentage of subjects who initiate such therapy will be calculated.
Percentage of subjects that initiate a standardized low key intervention | baseline
  All subjects will be offered the participation in a low key intervention as described in subproject two. The percentage of patients that accept and initiate this intervention will be calculated.
Percentage of subjects that participate in diagnostic procedures. | baseline
  Subjects will be offered a diagnostic liver ultrasound, sleep apnea screening, orthopedic screening, and an array of questionnaires to assess somatic- and psychiatric co-morbidities, psycho-social situation and health related quality of life. The percentage of subjects that comply with these diagnostic procedures beyond the initial visit will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Wabitsch, Prof. Dr. med., Study Chair — University of Ulm; Susanna Wiegand, Dr. med., Principal Investigator — Charite University, Berlin, Germany; Thomas Reinehr, Prof. Dr. med., Principal Investigator — University of Witten/Herdecke; Johannes Hebebrand, Prof. Dr. med., Principal Investigator — Universität Duisburg-Essen; Wieland Kiess, Prof. Dr. med., Principal Investigator — University of Leipzig; Reinhard Holl, Prof. Dr. med., Principal Investigator — University of Ulm; Anja Moss, Dr. biol. hum., Study Director — University of Ulm; Belinda S Lennerz, Dr. med., Study Director — University of Ulm; Julia von Schnurbein, Dr. med., Study Director — University of Ulm
Locations (5):
- Germany (5):
  - Ambulatory Obesity Program, Charité University, Berlin, Berlin
  - Vestische Kinderklinik, University of Witten/Herdecke, Datteln
  - University Duisburg-Essen, Essen
  - University Hospital Leipzig, Leipzig
  - Dept for Pediatrics and Adolescent Medicine, University of Ulm: Interdisciplinary obesity clinic, Ulm

REFERENCES:
- [Derived] Felix J, Stark R, Teuner C, Leidl R, Lennerz B, Brandt S, von Schnurbein J, Moss A, Bollow E, Sergeyev E, Muhlig Y, Wiegand S, Holl RW, Reinehr T, Kiess W, Scherag A, Hebebrand J, Wabitsch M, Holle R. Health related quality of life associated with extreme obesity in adolescents - results from the baseline evaluation of the YES-study. Health Qual Life Outcomes. 2020 Mar 5;18(1):58. doi: 10.1186/s12955-020-01309-z. PMID 32138734
- [Derived] Wabitsch M, Moss A, Reinehr T, Wiegand S, Kiess W, Scherag A, Holl R, Holle R, Hebebrand J. Medical and psychosocial implications of adolescent extreme obesity - acceptance and effects of structured care, short: Youth with Extreme Obesity Study (YES). BMC Public Health. 2013 Aug 29;13:789. doi: 10.1186/1471-2458-13-789. PMID 23987123
- See also: study homepage — http://www.adipositasforschung-ulm.de/index.php?id=69